CLINICAL TRIAL: NCT04612179
Title: Post-Market Registry to Evaluate the Safety and Efficacy of the The SUPRAFLEX CRUZ™ Sirolimus Eluting Coronary Stent System in the Treatment of an Octo- and Nonagenerian All-Comer Patient Cohort With Coronary Artery Disease - the Cruz Senior Study
Status: Completed | Type: Observational
Sponsor: IHF GmbH - Institut für Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: Cruz-Senior
Record Dates: First submitted 2020-10-30; First posted 2020-11-02 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Coronary Disease
Keywords: CAD; PCI; Cruz Stent; CCS; NSTE-ACS
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All Comer Patients: All-comer patients (≥80 years) affected by acute coronary syn-drome (NSTE-ACS), stabile angina, or silent angina, who qualify for percutaneous coronary intervention (PCI) according to ESC-treatment guidelines and physicians' clinical routine estimation.
  Interventions: Device: The SUPRAFLEX CRUZ™ Sirolimus eluting coronary stent system

INTERVENTIONS:
Device: The SUPRAFLEX CRUZ™ Sirolimus eluting coronary stent system — Investigational device: SUPRAFLEX CRUZ™ Sirolimus eluting Coronary Stent System The SUPRAFLEX CRUZ™ Sirolimus eluting coronary stent system consists of a balloon ex-pandable Sirolimus eluting stent, premounted on a stent delivery system. The active pharmaceutical ingredient in the SUPRAFLEX CRUZ™ Sirolimus eluting coronary stent is Sirolimus (also known as Rapamycin).
  The SUPRAFLEX CRUZ™ Sirolimus eluting coronary stent system is indicated for improving coronary luminal diameter in patients with symptomatic Ischemic heart disease due to discrete de-novo stenotic lesions and in-stent restenotic lesions in native coronary arter-ies with a reference vessel diameter of 2.00 mm to 4.50 mm.

SUMMARY:
Prospective, multi-centre, open-label, single-armed, non-interventional observational clinical investigation designed to enrol 2000 octo- and nonagenerian all-comer patients with coro-nary artery disease in up to 37 sites in Germany, Switzerland and Austria. Patients underwent PCI using at least one Supraflex Cruz Sirolimus Eluting stent as per current practice and will be followed up for 12 months.

DETAILED DESCRIPTION:
This is a prospective, multicentre, open-label, single-armed, non-interventional observa-tional clinical investigation in aged patients (≥80 years) undergoing PCI using at least one Supraflex sirolimus eluting stent as per current practice. The registry is an observational study and patient's participation in this study has no impact on his or her indication for treatment, diagnostics, or therapy. Subjects are supposed to be treated according to cur-rent guidelines and the site's internal directives.

Inclusion in the registry is completely independent of the medical treatment. All products used for the medical treatment should be administered as stated in their SmPCs (Sum-mary of Product Characteristics) and/or Instructions for Use (IFU). Treatment pattern and treatment initiation, continuation, or changes are solely at the discretion of the physician and the patient. There will be no attempt to influence the treatment patterns of any indi-vidual treating physician. All drug subscriptions applied will be in the usual standard of care. Participation in the registry will in no way influence payment or reimbursement for any treatment received by subjects during the study.

The study will be conducted about 37 sites in Germany, Switzerland and Austria and 2000 subjects will be included. A total study duration of about 39 months is assumed, of which about 18 months account for enrolment and 12 months for the follow-up.

Eligible are all patients with chronic- (CCS) or acute- Non-ST-elevation coronary syndrome (NSTE-ACS) and target lesion suitable for PCI with drug-eluting stent (see section 6.3 for detailed eligibility criteria) undergoing PCI using at least one SUPRAFLEX CRUZ™ Sirolimus eluting coronary stent system as per current practice, who will visit consecutively a partici-pating investigation site. It is planned to enroll about 2000 patients in total.

Following discharge, patients will be treated according to clinical routine/guidelines. Hence, no study-specific pre-planned procedures will be performed.

To assess the primary endpoint, all patients will receive telephone calls at 6 and 12 months following index procedure and will be interviewed by means of a standardized patient interview by the investigation sites.

On-site monitoring will be performed (about 1.5 visits per site; risk-based approach). Dur-ing on-site monitoring, the monitor will verify patient informed consent documentation and perform source data verification against the patient's medical records. In addition, an attempt will be made to check the consecutiveness of patient enrolment at the site, fully respecting privacy and personal data of subjects who are not enrolled in the registry and consequently have not given informed consent.

Data will be captured at three time points:

* Baseline (e.g. site and patient characteristics, index procedure, events, etc.),
* 6-months FU (e.g. vital status, endpoint-related events, quality of life, adverse events, etc.) and
* 12-months FU (e.g. vital status, endpoint-related events, quality of life, adverse events, etc.)

ELIGIBILITY:
Inclusion Criteria:

1. Written consent received from the patient or a legal repre-sentative after the information has been provided.
2. ≥ 80 years of age.
3. De-novo or re-stenotic significant stenosis in at least one cor-onary vessel.
4. Patients with NSTE-ACS, unstable angina, stable angina, silent ischemia (no limitation of the number of treated lesions and vessels: planned staged procedures are allowed within 3 months using Supraflex Cruz only).
5. Target lesion suitable for PCI with SUPRAFLEX CRUZ™ Siroli-mus eluting coronary stent system with diameter between 2.0 and 4.5 mm
6. Total lesion length should be from 6-120 mm

Exclusion Criteria:

1. Patients with ST-elevation myocardial infarction (STE-ACS)
2. Hemodynamic instability or cardiogenic shock
3. Known hypersensitivity or contraindication to any component of the study stent or the eluting drug, to media contrast, to dual antiplatelet therapy (DAPT) medication required by cur-rent practice
4. Any co-morbid condition with life expectancy < 1 year or that may result in protocol non-compliance
5. Patients who are participating in another drug or device inves-tigational study, which has not reached its primary endpoint
6. Patients under judicial protection, tutorship or curatorship

Ages: 80 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All-comer patients (≥80 years) affected by acute coronary syn-drome (NSTE-ACS), stabile angina, or silent angina, who qualify for percutaneous coronary intervention (PCI) according to ESC-treatment guidelines and physicians' clinical routine estimation.
Sampling Method: Non-Probability Sample
Enrollment: 2017 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Device Oriented Composite Endpoint | 12 month
  Device Oriented Composite Endpoint (DOCE as per ARC2) at 12 months defined as compo-site of cardiovascular death, myocardial infarction (MI) not clearly attributable to a non-target vessel and clinically driven target lesion revascularization (TLR)

SECONDARY OUTCOMES:
All death | 6 and 12 month
  All death, cardiovascular death and non-cardiovascular death rate
All MI rate | 6 and 12 month
  All MI rate at 6 months and 12 months
Rate of TV-MI and MI not | 6 and 12 month
  Rate of TV-MI and MI not clearly attributable to non-target vessel at 6 months and at 12 months
Clinically indicated TLR | 6 and 12 month
  Clinically indicated TLR rate at 6 months and 12 months.
All TLR rate | 6 months and at 12 months.
  All TLR rate at 6 months and at 12 months.
Target Vessel Revascularization (TVR | 6 months and at 12 months.
  All Target Vessel Revascularization (TVR) rate at 6 months and at 12 months.
revascularization rate | 6 months and at 12 months.
  All revascularization rate at 6 months and at 12 months.
Stent Thrombosis | 6 months and at 12 months
  Stent Thrombosis rate at 6 months and at 12 months (ARC2).
Device success | 12 month
  Device success defined as deployment of the stents without system failure or device-related complication
Lesion success | 12 month
  Lesion success defined as the attainment of < 50 % residual stenosis of the target le-sions post-PCI.
Procedure success | 12 month
  Procedure success defined as all lesion successfully treated without the occurrence of DOCE during the hospital stay.
Major Bleeding | 12 month
  Major Bleeding (BARC 3 to 5).
SAQ | 6 months
  Seattle Angina Questionnaire (SAQ) at 6 months
Quality of life PROMIS | 6- and 12-months
  Quality of life at 6- and 12-months as measured by PROMIS-29 questionnaire
Geriatric Assessment - Bartel Index | baseline
  Geriatric Assessment Questionnaire: Barthel-Index
Geriatric Assessment - Times up and Go Test | baseline
  Geriatric Assessment Questionnaire: Timed up - and Go Test
Geriatric Assessment - Minimal Mental Status Test | baseline
  Geriatric Assessment Questionnaire: Minimal Mental Status Test
Geriatric Assessment - G8 Questionnaire | baseline
  Geriatric Assessment Questionnaire: G8 Questionnaire
Geriatric Assessment - General Living conditions | baseline
  Geriatric Assessment Questionnaire: general living condition

CONTACTS AND LOCATIONS:
Overall Officials: David M Leistner, Prof, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided